CLINICAL TRIAL: NCT05482984
Title: Effects of Video-recorded Role-play and Guided Reflection on Nursing Student Empathy, Caring Behavior, and Competence: A Two-group Pretest-posttest Study
Brief Title: Effects of Video-recorded Role-play and Guided Reflection on Nursing Student Empathy, Caring Behavior, and Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, Researchers, Mackay Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21MMHIS315e
Record Dates: First submitted 2022-07-16; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Competence
Keywords: empathy; caring behavior; nursing competence; role play; reflection

STUDY DESIGN:
Intervention Model Description: The investigators used a two-group pretest and post-test quasi-experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lectures with video-recorded role-play and guided reflection (Experimental): The learning method used with the intervention group was role-playing with videos and guided reflection.
  Interventions: Other: video-recorded role-play and guided reflection
- Lectures without video-recorded role-play and guided reflection (No Intervention): The control group was exposed to classroom lectures without video-recorded role-play and guided reflection.

INTERVENTIONS:
Other: video-recorded role-play and guided reflection — The experimental group was divided into 6 teams. Before the course, the teacher in charge and each group developed six scenarios: restraint, suicidal intent, respiratory distress, chronic heart failure, medication refusal, and accidental amputation. The researcher guided each group to write scripts about the clinical situations (30 minutes), create role-play videos (50 minutes), and share literature that was helpful in understanding this context (30 minutes). Each student played a role in the filming process. The final film was viewed by all the students during class. Each live class session was 50 minutes in length, with one session per week for 6 weeks. All students were asked to attend six video-viewing sessions and participate in a reflective discussion.
  Arms: Lectures with video-recorded role-play and guided reflection

SUMMARY:
Objectives: To examine the differences in nursing student empathy, caring behaviour, and competence between the experimental and control groups before and after educational intervention, and to predict the factors affecting their core competencies.

DETAILED DESCRIPTION:
Design: The investigators used a two-group pretest and post-test quasi-experimental design.

Setting: The experiment was conducted at a college in northern Taiwan. Participants: First-year nursing students from medical schools in Taiwan participated in our study.

Methods: Data were collected between March and May 2022. The learning method used with the intervention group was role-playing with videos and guided reflection. The control group was exposed to classroom lectures without video-recorded role-play and guided reflection. Empathy, caring behaviour, and competence were measured using the Jefferson Scale of Empathy- Healthcare Providers, the Caring Behaviours Scale, and the Nursing Student Competence Scale.

ELIGIBILITY:
Inclusion Criteria:

* (1) Students who were first-year nursing students at college,
* (2) could communicate using Mandarin or Taiwanese,
* (3) were willing to participate in this study and agreed to cooperate with the completion of the questionnaire.

Exclusion Criteria:

* deafness or a diagnosis of cognitive disorder according to various information sources, such as school health information and notification from parents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Nursing Student Competence Scale | Baseline data were collected 1 week prior to the intervention study. The second data were collected 1 week after the implementation of the intervention and up to 2 weeks.
  The Nursing Student Competence Scale was used to measure students' nursing competence (Huang et al., 2022). Total scale scores ranged from 30 to 150. Higher scores indicate better nursing competence.

SECONDARY OUTCOMES:
Change from Jefferson Scale of Empathy- Healthcare Providers | Baseline data were collected 1 week prior to the intervention study. The second data were collected 1 week after the implementation of the intervention and up to 2 weeks.
  Empathy was measured using the Chinese version of the Jefferson Scale of Empathy- Healthcare Providers, developed based on a literature review (Cheng et al., 2011). Total scale scores ranged from 20 to 140. Higher scores indicate more positive empathy.
Change from Caring Behaviours Scale | Baseline data were collected 1 week prior to the intervention study. The second data were collected 1 week after the implementation of the intervention and up to 2 weeks.
  The Caring Behaviours Scale, with 27 items, was used to measure students' caring behaviours (Lin, 2001; Pai et al., 2013). Total scale scores ranged from 27 to 108. Higher scores indicate a greater frequency of caring behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Miauh Huang, PhD, Principal Investigator — Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No